CLINICAL TRIAL: NCT07039175
Title: A Low-Cost, High-Access Intervention to Increase Intention to Change Alcohol/Tobacco Use Among Reticent Veterans Who Are Non-Responders to Brief Advice at High Risk Due to Chronic Conditions
Brief Title: Intervention to Increase Intention to Change Alcohol/Tobacco Use in Veterans With Chronic Disease
Acronym: MINDSET
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 23-170; 1IOHX003901 (Other Grant/Funding Number: VA Health Services Research)
Record Dates: First submitted 2025-06-13; First posted 2025-06-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Tobacco Smoking; Alcohol-Related Disorders
Keywords: Chronic Disease; Smoking; Drinking, Alcohol; Cardiovascular Risk; Health Behavior; Medicine, Behavioral; telehealth
MeSH Terms: conditions — Tobacco Smoking; Alcohol-Related Disorders; Chronic Disease; Smoking; Alcohol Drinking; Health Behavior; Behavior | interventions — Stress Mindset Measure; Self-Management; Educational Status

STUDY DESIGN:
Intervention Model Description: Participants recruited from VAs across the country will be randomized to receive usual care + MINDSET or usual care alone.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blinded to the condition of the Veteran at all assessment time points.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MINDSET+UC (Experimental): Within one month following a standard primary care appointment (which comprises usual care; UC), Veterans in this condition will receive the MINDSET intervention which consists of: a behavior-change model informed mailed informational packet with tailored health information regarding the impacts of smoking/drinking on chronic disease and the benefits of stopping, followed by a brief motivational telephone booster call from a behavioral health provider.
  Interventions: Behavioral: MINDSET
- Usual Care (Active Comparator): All Veterans in this study will have a primary care appointment during which their primary care team will administer whatever tobacco/alcohol use assessment and intervention they typically would.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: MINDSET — A behavior-change model informed mailed informational packet with tailored health information regarding the impacts of smoking/drinking on chronic disease and the benefits of stopping, followed by a brief motivational telephone booster call from a behavioral health provider.
  Other Names: Motivational INtervention Designed for Self-management and EducaTion
  Arms: MINDSET+UC
Other: Usual Care — All Veterans involved in this study will have a standard primary care (PC) appointment, which may include conversations/interventions related to drinking and smoking. This appointment is not controlled by the study team and we cannot comment on the extent to which smoking/drinking will or will not be discussed in the primary care appointment but we imagine this can range from no discussion/intervention at all to extensive conversations with the provision of medications, brief advice, etc.
  Other Names: UC
  Arms: Usual Care

SUMMARY:
Many Veterans who have chronic conditions like cardiovascular disease or diabetes smoke or drink too much alcohol, which can worsen the condition. Veterans are asked yearly about drinking/smoking and providers provide a brief advice discussion focused on behavior change. However, many Veterans continue to drink or smoke, and are often not interested in higher-intensity, change-based referrals. The investigators recently piloted MINDSET, an intervention that fills this gap. MINDSET is a proactive, population-based intervention that uses a mailed packet with tailored education about how drinking/smoking relate to the Veteran's condition (heart conditions and/or diabetes), followed by a brief motivational call. The investigators will test MINDSET's effectiveness versus usual primary care on outcomes including intention to change and substance use and evaluate the relationships between these and other variables over time.

DETAILED DESCRIPTION:
Background: Chronic diseases are prevalent, costly, and have been linked to increased risk of mortality and morbidity in Veterans. Hazardous alcohol use and cigarette smoking can significantly exacerbate these negative consequences for Veterans. To help mitigate risk, VHA primary care health initiatives have prioritized hazardous alcohol use and cigarette smoking and have mandated that patients be annually screened and receive a brief intervention (primary care intervention delivered by the patient-aligned care team; PACT) if positive. However, many Veterans continue to smoke and/or hazardously drink. Current VHA treatment options do not meet the needs of these reticent Veterans. Motivational Intervention Designed for Self-management and EducaTion (MINDSET) is an evidence-based, remote, low-resource intervention that uses a motivational approach to increase change intentions within the context of their chronic disease.

Significance: Most healthcare costs come from Veterans with chronic diseases (e.g., cardiovascular disease; CVD), which are worsened by hazardous alcohol use and smoking. This research addresses multiple VHA priorities through its focus on increasing access to care for a subgroup of reticent Veterans with chronic disease. MINDSET's integrated focus on smoking and hazardous drinking in the context of chronic disease management aligns with Veteran's priorities, and diabetes and CVD were a top ranked health concern by Veterans. This work is also very well aligned with several HSR&D Priorities, including Complex Chronic Disease Management, Mental & Behavioral Health, Women's Health, Aging, and Access to Care.

Innovation & Impact: MINDSET's design, which recognizes the competing demands within medical settings, intentionally utilizes universal and accessible dissemination methods (e.g., mail and telephone) to decrease burden while increasing reach and impact. This study uniquely fills a gap in VHA and HSR&D research as there are no evidence-based interventions tailored for this subgroup of reticent Veterans who smoke and/or drink above recommended limits and have co-occurring CVD, cardiac risk factors, and/or diabetes. The impact potential is high, as moving this subgroup of reticent Veterans toward changing smoking/hazardous drinking will dramatically decrease their health risks and healthcare costs.

Specific Aims: The proposed work will evaluate MINDSET+usual care (UC) in comparison to UC alone (brief primary care advice) on precursors to change (i.e., behavioral control, intention to change), and substance consumption.

Methodology: The investigators will conduct a type 1 hybrid effectiveness-implementation RCT, where enrolled Veterans will be randomized to either the intervention condition UC (i.e., primary care brief advice) alone or (usual care [UC]+MINDSET). Assessments will occur every 4 weeks, with comprehensive assessments every 3 months for one year. The investigators will utilize a stratified block randomization method based on whether Veterans report only smoking, only hazardously drinking, or both. The investigator's primary outcome will assess participants' intention to change each behavior separately, and a total summed score across items divided by the number of items endorsed (based on behaviors engaged in) will be utilized to summarize their overall intention to change. It is important to note that Veterans will be recruited nationally for this fully telehealth-based study.

Next Steps/Implementation: If MINDSET is effective, additional implementation research/efforts will be proposed.

ELIGIBILITY:
Inclusion Criteria:

* an active diagnosis of diabetes, cardiovascular disease (CVD), or a cardiovascular risk factor (hypertension {HTN}, hyperlipidemia {HLD}) AND signs of reticence to change their smoking and/or alcohol use as evidenced by the two consecutive prior screens being positive for hazardous (e.g., Alcohol Use Disorders Test-Consumption [AUDC], and/or smoking (I.e., whether they are a current smoker or not).
* Confirmation of smoking and/or drinking status during telephone screening (e.g., Alcohol Use Disorders Test-Consumption [AUDC], and/or smoking (I.e., whether they are a current smoker or not).
* Veteran
* Age 18 years
* utilize VA for medical care more than 1 time per year
* are due to complete their smoking/alcohol use screen in approximately 3 months (to ensure they will likely receive UC during intervention period)
* a scheduled PC appointment within the intervention period.

Exclusion Criteria:

* dementia or severe cognitive impairment per Problem List
* significant visual impairment per Problem List
* Other Exclusion criteria assessed by study staff during screening/self-report are:

  * inability to communicate or read in English;
  * Hearing impairment; and
  * cognitive impairment or screening for cognitive impairment (>=weighted score of 10 on Blessed screener).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Theory of Planned Behavior Intention subscale | Baseline, 4-weeks, 8-weeks, 12-weeks, 16-weeks, 20-weeks, 24-weeks, 28-weeks, 32-weeks, 36-weeks, 40-weeks, 44-weeks, 48-weeks
  3 items regarding intention to change measured on a 7-point Likert-type scale from (1) very unlikely to (7) very likely.
Readiness to Change Ruler | Baseline, 4-weeks, 8-weeks, 12-weeks, 16-weeks, 20-weeks, 24-weeks, 28-weeks, 32-weeks, 36-weeks, 40-weeks, 44-weeks, 48-weeks
  A one-item 11-point (0-10) ruler with the following anchors: "I never think about my drinking/smoking" at 0 to "I now drink/smoke less than before" at 10
Theory of Planned Behavior Perceived Behavioral Control Subscale | Baseline, 4-weeks, 8-weeks, 12-weeks, 16-weeks, 20-weeks, 24-weeks, 28-weeks, 32-weeks, 36-weeks, 40-weeks, 44-weeks, 48-weeks
  4 items measured on a 1-7 point Likert-type scale. The four items include two related to self-efficacy and two to controllability, as recommended by guidelines for developing TBP-related measurements.

SECONDARY OUTCOMES:
Timeline Followback | Baseline, 12-weeks, 24-weeks, 36-weeks, 48-weeks
  A verbal/guided measure that guides Veterans Veterans through the last 90 days reporting how many drinks or cigarettes they had each day.
Theory of Planned Behavior Action Planning subscale | Baseline, 12-weeks, 24-weeks, 36-weeks, 48-weeks
  4 items (e.g., I have been thinking about when I'm going to change) that measure planning/action behaviors toward change based on TBP rated on a 7-point Likert-type scale from (1) completely wrong to (7) complete correct.
Theory of Planned Behavior Quitting Behaviors subscale | Baseline, 12-weeks, 24-weeks, 36-weeks, 48-weeks
  3 dichotomous face-valid questions to assess the participants quitting/change behaviors (e.g., "I have quit") on a yes-no scale
Readiness to Access Help scale plus Help-Seeking for Alcohol-Related Problems Scale | Baseline, 12-weeks, 24-weeks, 36-weeks, 48-weeks
  6-items that will be used to assess any help seeking behaviors (e.g., accessing self-help resources) that has already occurred on a 11-point Likert-scale. Two additional items adapted from the Help-Seeking for Alcohol-Related Problems in College Students Scale106 will be included attending group meetings and calling a counselor or doctor.

OTHER OUTCOMES:
Client Satisfaction Questionnaire | 24-week post assessment only
  8-item self-report questionnaire on patient satisfaction with medical and mental health interventions, with higher scores indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Christina Gass, PhD, Principal Investigator — VA Western New York Healthcare System, Buffalo, NY; Jennifer S Funderburk, PhD, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY
Locations (1):
- VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No